CLINICAL TRIAL: NCT01907477
Title: Identification of Serum and/or Plasma Biomarkers for the Diagnosis Prognosis and/or Prediction of Invasive Mycosis in Neutropenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dalle PHRC IR 2009
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2013-07

CONDITIONS: Neutropenic Patients

ARMS (1):
- neutropenic patients (Other)
  Interventions: Other: Samples taken at the clinical hematology unit

INTERVENTIONS:
Other: Samples taken at the clinical hematology unit

SUMMARY:
The aim of the present work is to study the protein expressions profiles of neutropenic patients (with a high risk of invasive mycosis) who developed - versus who did not develop invasive mycosis (principally aspergillosis and candidosis) in order to identify biomarkers for the diagnosis, prognosis and /or prediction of invasive mycosis.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with malignant haemopathy who received chemotherapy likely to lead to severe neutropenia (PN<500/mm3) for a foreseeable period of 10 days.
* Patients aged 14 years or older (no upper age limit)
* Patients with malignant haemopathy who received an autologous marrow graft.
* Patients with severe idiopathic medullar aplasia (PN<500/mm3) who need to be hospitalised for at least 10 days consecutively (with or without immunosuppressant treatment).
* Patients who have provided written informed consent to participate in this study.

Exclusion Criteria:

* Patients who received an allograft of marrow or hematopoietic stem cell transplant (given that these patients carry a risk of aspergillosis, which in most cases appears after medullar recovery, they will not be included in the study).
* Patients who received an autologous hematopoietic stem cell transplant (given that the duration of the neutropenia is often less than 10 days).
* Patients who do not meet the inclusion criteria
* Persons not covered by the national Health Insurance Agency

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
the variability of protein profiles | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France